CLINICAL TRIAL: NCT02625298
Title: Use of Mineral Trioxide Aggregate in the Treatment of Traumatized Permanent Teeth With Necrotic Pulps and Chronic Periapical Lesions
Brief Title: Use of Mineral Trioxide Aggregate in the Treatment of Traumatized Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association of Paediatric and Preventive Dentists of Serbia (Other)
Responsible Party: Principal Investigator, Dejan Markovic, Professor, Association of Paediatric and Preventive Dentists of Serbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001-12
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-07

CONDITIONS: Periapical Diseases
Keywords: periapical diseases; dental injuries; MTA
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ProRoot MTA (Experimental): Traumatized permanent teeth obturated with ProRoot MTA after root canal treatment
  Interventions: Device: ProRoot MTA
- MTA+ Cercamed (Experimental): Traumatized permanent teeth obturated with MTA+ Cerkamed after root canal treatment
  Interventions: Device: MTA+ Cerkamed

INTERVENTIONS:
Device: ProRoot MTA — Apical thirds of the root canals obturated with ProRoot MTA (Dentsply Tulsa Dental Specialties, Tulsa, OK USA).
  Arms: ProRoot MTA
Device: MTA+ Cerkamed — Apical thirds of the root canals obturated with MTA + (Cerkamed, Stalowa Wola, Poland).
  Arms: MTA+ Cercamed

SUMMARY:
Traumatic tooth injuries are common in children and adolescents, and often result in pulpal necrosis and the development of periapical lesions. Treatment of traumatized teeth with endodontic complications depends on the type of injury, number of injured teeth, root development and patient cooperation, which altogether will create a challenge and dictate the treatment plan for the dentist. The purpose of this study was to assess the effectiveness of non-surgical root canal procedures in traumatized permanent teeth with necrotic pulps and chronic periapical lesions using a tri-antibiotic paste and calcium-hydroxide as intracanal medications and two different mineral trioxide aggregate (MTA) products for definitive obturation.

DETAILED DESCRIPTION:
Root canal procedures will be performed on single-rooted traumatized permanent teeth (both with mature and immature root development) with necrotic pulps and periaoical lesions. Following access opening in each tooth, the root canals will be gently debrided with a crown-down manual technique using K-files according to the radiographically determined working lengths; irrigation with saline was used in all cases. K-files will be only used to remove the necrotic tissue and the softened predentinal layer without excessive removal of mineralized dentin, as this may have further weaken already thin walls of the root canals, particularly those with immature apical development. Subsequently, a reshaping of the canal system, followed by a minor curettage of the periapical area through the canal using barbed broaches will be made in order to partially destruct the periapical lesion and provoke bleeding. Final irrigation will be performed using 2% NaOCl (Chloraxid, Cerkamed, Stalowa Wola-Poland), 0.2% solution of chlorhexidine-digluconate (Curasept 220, Curadent Swiss GmbH, Kriens-Switzerland) and 40% citric acid solution (40% Citric acid, Cerkamed, Stalowa Wola, Poland). The canals will be then dried with sterile paper points and filled with triple-antibiotics paste using a lentula, for a period of seven days. Following this initial disinfection, calcium-hydroxide paste will be placed into the root canals for at least four weeks, for a maximum of six weeks (UltraCal XS, Ultradent Products Inc., South Jordan, UT USA). Apical thirds of the root canals will be obturated either with ProRoot MTA (Dentsply Tulsa Dental Specialties, Tulsa, OK USA) or MTA+ Cerkamed (Cerkamed, Stalowa Wola, Poland) by forming an apical plug of 3-5 mm of thickness. The correct placement of the apical plug will be assessed radiographically, and the moist cotton pellet was left in the root canal. The next day, the rest of the canal space will be filled with a sealer (Acroseal, Septodont, Saint-Maur des Frosses-France) and gutta-percha points (Guttapercha, VDW GmbH, Munich-Germany) using a lateral compaction technique. Coronal parts of root canal systems will be sealed using glass-ionomer cement (Fuji IX, GC Int., Tokyo, Japan) with a minimum thickness of 1.5-2 mm. The teeth will be restored using composite material (Gradia Direct, GC Int., Tokyo, Japan). Two dentists with many years of clinical experience, and using identical, predetermined treatment protocols will perform all treatments.

The positive clinical outcome will comprise of absence of spontaneous or provoked pain, no discomfort during chewing, no numbness or tenderness to percussion and/or palpation, no altered tooth mobility, tooth crown discoloration or abscess and/or sinus tract. Radiological assessment of the outcomes will be performed according to the analysis of post treatment radiographs (initial, baseline, 3, 6, 12, and 24-months subsequent to obturation) after being photographed using a digital camera Kodak EasyShare Max (Z990) with millimetre measurer in order to obtain interpretation of sizes of periapical lesions during conversion of pixels in mm2 by digital data processing in Adobe Photoshop CS software.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient
* Non-vital tooth with chronic periapical lesions
* Restorable tooth
* No horizontal or vertical root fractures
* No root resorption

Exclusion Criteria:

* Unrestorable tooth
* Horizontal or vertical root fractures
* Root resorption

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study involved twenty-four patients, 11 males (45.8%) and 13 females (54.2%) (mean age 13.30±2.83), who came to the University Clinic, due to spontaneous or provoked pain, discomfort during chewing, numbness, and observed swelling.
Pre-assignment Details: Based on patient's subjective symptoms, clinical examination, vitality testing and analysis of periapical radiograph, the acute exacerbation of a necrotic pulp with chronic apical periodontitis was diagnosed. If the teeth were unrestorable or with signs of horizontal or vertical root fractures or root resorption, they were excluded from this study.
Period: Overall Study
Arm/Group | ProRoot MTA | MTA+ Cercamed
Started | 11 | 13
Completed | 10 | 13
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: tooth
Groups:
- Total: Total of all reporting groups
Arm/Group | ProRoot MTA | MTA+ Cercamed | Total
Number analyzed (Participants) | 11 | 13 | 24
Number analyzed (tooth) | 14 | 13 | 27
Age, Categorical [Count of Units; unit: tooth]
  <=18 years | 14 | 13 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: tooth]
  Serbia | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Changes Between Initial and Post Treatment Dimensions of Periapical Lesions
Description: Changes in the dimensions of periapical lesions will be performed according to the analysis of initial and post treatment radiographs (baseline, 3, 6, 12, and 24-months subsequent to obturation) after being photographed using a digital camera Kodak EasyShare Max (Z990) with millimetre measurer in order to obtain interpretation of sizes of periapical lesions during conversion of pixels in mm2 by digital data processing in Adobe Photoshop CS software. Sucessful radiographic assessment will include decrease in size of the periapical lesion at the recall time of 24 months.
Time Frame: baseline, 3, 6, 12 and 24 months
Measure: Mean (Standard Deviation); unit: square millimeters
Units Other Than Participants: tooth
Arm/Group | ProRoot MTA | MTA+ Cercamed
Number analyzed (Participants) | 11 | 13
Number analyzed (tooth) | 14 | 13
square millimeters
  Initial | 37.34 (0.63) | 34.04 (0.34)
  Baseline | 16.20 (0.21) | 17.54 (0.75)
  3 months | 12.74 (0.19) | 12.01 (0.34)
  6 months | 11.59 (0.25) | 7.86 (0.23)
  12 months | 8.38 (0.10) | 4.85 (0.24)
  24 months | 2.99 (0.10) | 2.48 (0.10)
Statistical Analysis 1: Comparison: ProRoot MTA vs MTA+ Cercamed; Test type: Other; p < 0.01, Mixed Models Analysis

2. Secondary Outcome: Presence of Clinical Symptoms
Description: Clinical examination will be used to assess the presence of spontaneous or provoked pain, discomfort during chewing, numbness or tenderness to percussion and/or palpation, altered tooth mobility, tooth crown discoloration or abscess and/or sinus tract.
Time Frame: baseline
Measure: Number; unit: participants
Arm/Group | ProRoot MTA | MTA+ Cercamed
Number analyzed (Participants) | 11 | 13
participants
  spontaneous or provoked pain | 5 | 5
  discomfort during chewing | 8 | 6
  numbness | 3 | 1
  tenderness to percussion and/or palpation | 2 | 2
  altered tooth mobility | 2 | 1
  tooth crown discoloration | 1 | 1
  abscess and/or sinus tract | 1 | 0

ADVERSE EVENTS:
Description: Serious Adverse Events were not monitored/assessed.
Arm/Group | ProRoot MTA | MTA+ Cercamed
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No